CLINICAL TRIAL: NCT02466607
Title: Study of Stimulus Parameters in Flicker Electroretinogram (ERG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LKC Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Purpose: Basic Science
Other Study IDs: SAIRB-15-0017
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Retinopathy
Keywords: Retinal function
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RETeval color flicker ERG (Other): Compare implicit times and amplitudes of electroretinograms obtained from series of color flashes to those obtained from white flashes.
  Interventions: Device: RETeval color flicker ERG
- RETeval dilated versus un-dilated flicker ERG (Other): Compare implicit times and amplitudes of ERGs obtained from cd/m2/sec stimulation (used with dilated pupils) to those obtained from troland stimulation (used with un-dilated pupils).
  Interventions: Device: RETeval dilated versus un-dilated flicker ERG; Other: pupil dilation

INTERVENTIONS:
Device: RETeval color flicker ERG — Flicker ERGs obtained to 56 CIE 1931 (created by the International Commission on Illumination (CIE) in 1931) colors series. White flash of 0,33, 0,33 was used for comparison.
  Arms: RETeval color flicker ERG
Device: RETeval dilated versus un-dilated flicker ERG — Two series of white flashes: 3,0 cd/m2/sec and Trolands equivalent assuming 3,7 mm pupil size, delivered at 3 min interval over 30 min.
  Arms: RETeval dilated versus un-dilated flicker ERG
Other: pupil dilation — Pupil will be dilated using Proparacaine 0.5% and Tropicamide 0.5%
  Arms: RETeval dilated versus un-dilated flicker ERG

SUMMARY:
The electroretinogram (ERG) is a diagnostic test that measures the electrical activity generated by cells in the retina in response to a light stimulus. Typically, an ERG is recorded with white flash when the pupil is dilated. RETeval Visual Diagnostic Device (RETeval) generates an array of color flashes, which allows studying whether color flash would be a useful diagnostic tool.

Full pupil dilation is required to obtain a response from the whole retina. However, this requirement often limits a patient's flow in the clinic and increases the overall time patients spend at the eye practitioner. RETeval provides the possibility of recording ERGs in un-dilated pupils therefore making the whole exam easier and shorter. These results need to be compared to the classic, fully dilated ERG and evaluated for efficiency.

The purpose of this research study is to use the RETeval device to measure the eye's electrical response and how it changes with different stimuli such as changing flash color or pupil dilation.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers
* volunteers able to get their pupil fully dilated

Exclusion Criteria:

* pregnant women
* children
* subjects with
* light sensitivity
* photosensitive epilepsy
* allergies or sensitivity to pupil dilation ophthalmic solutions
* history of glaucoma
* cardiac dysrhythmia will not be invited to participate in this study.
* Pregnancy status, light sensitivity and photosensitive epilepsy will be based on volunteer's providing this information at the time of signing the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Flicker harmonic amplitude | up to 2 mnths
Flicker harmonic implicit time | up to 2 months
Flicker fundamental amplitude | up to 2 months
Flicker fundamental implicit time | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Olga Kraszewska, Ph.D., Principal Investigator — LKC Technologies
Locations (1):
- Wedgwood Optometry, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Davis CQ, Kraszewska O, Manning C. Constant luminance (cd.s/m2) versus constant retinal illuminance (Td.s) stimulation in flicker ERGs. Doc Ophthalmol. 2017 Apr;134(2):75-87. doi: 10.1007/s10633-017-9572-3. Epub 2017 Feb 3. PMID 28160194